CLINICAL TRIAL: NCT01475955
Title: A Phase II Study of Photodynamic Therapy With LEVULAN® Topical Solution + Blue Light Versus LEVULAN® Topical Solution Vehicle + Blue Light Using Spot and Broad Area Application and Incubation Times of 1, 2 and 3 Hours for the Treatment of Multiple Actinic Keratoses on the Face or Scalp
Brief Title: Short-incubation Levulan Photodynamic Therapy Versus Vehicle for Face/Scalp Actinic Keratosis (AK)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP0105
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Broad Area ALA 1-hour incubation (Experimental): Broad Area ALA 1-hour incubation
  Interventions: Drug: Broad Area ALA 1-hour incubation; Device: Blue Light Treatment
- Broad Area ALA 2-hour incubation (Experimental): Broad Area ALA 2-hour incubation
  Interventions: Drug: Broad Area ALA 2 hour incubation; Device: Blue Light Treatment
- Broad Area ALA 3-hour incubation (Experimental): Broad Area ALA 3-hour incubation
  Interventions: Drug: broad area ALA 3-hour incubation; Device: Blue Light Treatment
- Spot ALA 2-hour incubation (Experimental): Spot ALA 2-hour incubation
  Interventions: Drug: Spot ALA 2 hour incubation; Device: Blue Light Treatment
- Vehicle PDT (Placebo Comparator): VEH group will be randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH will be considered a single treatment group.
  Interventions: Drug: Vehicle PDT; Device: Blue Light Treatment

INTERVENTIONS:
Drug: Broad Area ALA 1-hour incubation — 20% ALA, broad area, 1 hour incubation
  Other Names: Levulan
  Arms: Broad Area ALA 1-hour incubation
Drug: Broad Area ALA 2 hour incubation — 20% ALA broad area 2-hour incubation
  Other Names: Levulan
  Arms: Broad Area ALA 2-hour incubation
Drug: broad area ALA 3-hour incubation — 20% ALA broad area 3 hour incubation
  Other Names: Levulan
  Arms: Broad Area ALA 3-hour incubation
Drug: Spot ALA 2 hour incubation — 20% ALA spot 2 hour incubation
  Other Names: Levulan
  Arms: Spot ALA 2-hour incubation
Drug: Vehicle PDT — Levulan Kerastick containing vehicle ingredients only.VEH group will be randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH will be considered a single treatment group.
  Arms: Vehicle PDT
Device: Blue Light Treatment — 10 J/cm2 blue light delivered at 10 mW/cm2
  Other Names: BLU-U

SUMMARY:
The purpose of this study is to determine if Levulan Photodynamic Therapy (PDT) is safe and effective in the treatment of actinic keratosis when applied to broad areas on the face and scalp for 1, 2 and 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* 6-20 Grade 1/2 AKs on the face or scalp
* a history of AK therapy within the treatment area at least twice in the two years prior to study entry

Exclusion Criteria:

* Pregnancy
* Grade 3 AKs or atypical AKs (e.g., AK > 1 cm2 in size) within the Treatment Area
* lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the Treatment Area
* plans to be exposed to artificial tanning devices or excessive sunlight during the trial
* Subject is immunosuppressed
* unsuccessful outcome from previous ALA-PDT therapy
* history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis
* skin pathology or condition which could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy
* skin pathology or condition that could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy
* any condition which would make it unsafe for the subject to participate in this research study
* currently enrolled in an investigational drug or device study
* has received an investigational drug or been treated with an investigational device within 30 days prior to the initiation of treatment
* known sensitivity to one or more of the vehicle components (ethyl alcohol, isopropyl alcohol, laureth 4, polyethylene glycol)
* Subject has;

  * an active herpes simplex infection OR
  * a history of 2 or more outbreaks within the past 12 months, in the Treatment Area
* use of the following topical preparations on the extremities to be treated:

  * Keratolytics including urea (greater than 5%), alpha hydroxyacids [e.g.glycolic acid, lactic acid, etc. greater than 5%], salicylic acid (greater than 2%) within 2 days of initiation of treatment.
  * Cryotherapy within 2 weeks of initiation of treatment
  * Retinoids, including tazarotene, adapalene, tretinoin, retinol, within 4 weeks of initiation of treatment.
  * Microdermabrasion, laser ablative treatments, ALA-PDT, chemical peels, 5-FU, diclofenac, imiquimod or other topical treatments for AK within 8 weeks of initiation of treatment.
  * Two or more ALA PDT treatments in the past 6 months
* use of systemic retinoid therapy within 6 months of initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Marcus, MD, PhD, Study Director — DUSA Pharmaceuticals, Inc.
Locations (13):
- United States (13):
  - UCSD Dermatology Perlman Ambulatory Clinic, La Jolla, California
  - Dermatology Research Associates, Los Angeles, California
  - Therapeutics Clinical Research, San Diego, California
  - Northwest Clinical Trials, Inc., Boise, Idaho
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Dermatology Research Center of Cincinnati, Cincinnati, Ohio
  - Oregon Medical Research Center, PC, Portland, Oregon
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - Suzanne Bruce and Associates, P.A.,The Center for Skin Research, Houston, Texas
  - Virginia Clinical Research Inc, Norfolk, Virginia

REFERENCES:
- [Derived] Piacquadio D, Berman B, Siegel DM, Bhatia N, Brocato J, Squittieri N, Pariser DM. Treatment Satisfaction and Acceptability of 20% Aminolevulinic Acid Photodynamic Therapy for the Treatment of Actinic Keratoses of the Face, Scalp, and Upper Extremities. J Clin Aesthet Dermatol. 2023 Dec;16(12):46-51. PMID 38125671

RESULTS

PARTICIPANT FLOW:
Groups:
- Broad Area ALA 1-hour + BLUE Light Treatment: Broad Area ALA 1-hour incubation : 20% ALA, broad area, 1 hour incubation, prior to BLUE light treatment at Visits 1 and 5
- Broad Area ALA 2-hour + BLUE Light Treatment: Broad Area ALA 2-hr incubation : 20% ALA broad area 2-hour incubation, prior to BLUE light treatment at Visits 1 and 5.
- Broad Area ALA 3-hour + BLUE Light Treatment: broad area ALA 3-hour incubation : 20% ALA broad area 3 hour incubation, prior to BLUE light treatment at Visits 1 and 5.
- Spot ALA 2-hour + BLUE Light Treatment: Spot application ALA 2 hour incubation : 20% ALA spot application 2 hour incubation, prior to BLUE light treatment at Visits 1 and 5.
- Vehicle + BLUE Light Treatment: Vehicle (VEH) group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment at Visits 1 and 5. Subjects receiving VEH were considered a single treatment group.
  Vehicle (VEH) Photodynamic Therapy (PDT) : Levulan Kerastick containing vehicle ingredients only.VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH were considered a single treatment group.
Period: Overall Study
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Started | 48 | 48 | 47 | 46 | 46
Completed | 47 | 48 | 44 | 46 | 46
Not Completed | 1 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Broad Area ALA 1-hour + BLUE Light Treatment: Broad Area ALA 1-hour incubation : 20% ALA, broad area, 1 hour incubation prior to BLUE light treatment at Visit 1 and Visit 5
- Broad Area ALA 2-hour + BLUE Light Treatment: Broad Area ALA 2-hr incubation : 20% ALA broad area 2-hour incubation prior to BLUE light treatment at Visit 1 and Visit 5
- Broad Area ALA 3-hour + BLUE Light Treatment: broad area ALA 3-hour incubation : 20% ALA broad area 3 hour incubation prior to BLUE light treatment at Visit 1 and Visit 5
- Spot ALA 2-hour + BLUE Light Treatment: Spot application ALA 2 hour incubation : 20% ALA spot application 2 hour incubation prior to BLUE light treatment at Visit 1 and Visit 5
- Vehicle (VEH) + BLUE Light Treatment: VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment at Visit 1 and Visit 5. Subjects receiving VEH were considered a single treatment group.
  Vehicle PDT : Levulan Kerastick containing vehicle ingredients only.VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH were considered a single treatment group.
- Total: Total of all reporting groups
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle (VEH) + BLUE Light Treatment | Total
Number analyzed (Participants) | 48 | 48 | 47 | 46 | 46 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.0) | 67.1 (9.4) | 66.4 (10.6) | 69.5 (9.7) | 68.4 (9.4) | 67.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 7 | 2 | 6 | 23
  Male | 45 | 43 | 40 | 44 | 40 | 212
Region of Enrollment [Number; unit: participants]
  United States | 48 | 48 | 47 | 46 | 46 | 235

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance Rate
Description: The proportion of subjects in each treatment group with a count of zero lesions in the Treatment Area
Time Frame: Week 12
Population: Intent to Treat (ITT) with last observation carried forward (LOCF) to impute missing data
Measure: Number; unit: participants
Groups:
- Vehicle + BLUE Light Treatment: VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment at Visits 1 and 5.. Subjects receiving VEH were considered a single treatment group.
  Vehicle PDT : Levulan Kerastick containing vehicle ingredients only.VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH were considered a single treatment group.
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants | 14 | 7 | 13 | 8 | 1
Statistical Analysis 1: Comparison: Broad Area ALA 1-hour + BLUE Light Treatment vs Broad Area ALA 2-hour + BLUE Light Treatment vs Broad Area ALA 3-hour + BLUE Light Treatment vs Spot ALA 2-hour + BLUE Light Treatment vs Vehicle + BLUE Light Treatment; Pearson chi-square; Test type: Superiority or Other; p = 0.0041, Chi-squared

2. Secondary Outcome: Complete Clearance Rate
Description: The proportion of subjects in each treatment group with a count of zero lesions in the Treatment Area
Time Frame: Week 4
Population: ITT LOCF
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants | 5 | 8 | 5 | 4 | 0

3. Secondary Outcome: Complete Clearance Rate
Description: The proportion of subjects in each treatment group with a count of zero lesions in the Treatment Area
Time Frame: Week 8
Measure: Number; unit: participants
Groups:
- Broad Area ALA 2-hour + BLUE Light Treatment: Broad Area ALA 2-hr incubation : 20% ALA broad area 2-hour incubation,prior to BLUE light treatment at Visits 1 and 5.
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants | 3 | 7 | 8 | 4 | 0

4. Secondary Outcome: Complete Clearance Rate
Description: the proportion of subjects in each treatment group with a count of zero lesions in the Treatment Area
Time Frame: Week 24
Measure: Number; unit: participants
Groups:
- Vehicle + BLUE Light Treatment: VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment at Visits 1 and 5. . Subjects receiving VEH were considered a single treatment group.
  Vehicle PDT : Levulan Kerastick containing vehicle ingredients only.VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH were considered a single treatment group.
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants | 11 | 3 | 12 | 2 | 1

5. Secondary Outcome: Partial Clearance Rate
Description: proportion of subjects with 75% or more reduction in the AK count in the Treatment Area as compared to baseline.
Time Frame: Baseline, Week 4
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants | 12 | 16 | 14 | 12 | 2

6. Secondary Outcome: Partial Clearance Rate
Description: proportion of subjects with 75% or more reduction in the AK count in the Treatment Area as compared to baseline.
Time Frame: Baseline, Week 8
Measure: Number; unit: participants
Groups:
- Vehicle + BLUE Light Treatment: VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment at Visits 1 and 5.. Subjects receiving VEH were considered a single treatment group.
  Vehicle PDT : Levulan Kerastick containing vehicle ingredients only.VEH group were randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH were considered a single treatment group.
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants | 10 | 13 | 15 | 13 | 1

7. Secondary Outcome: Partial Clearance Rate
Description: proportion of subjects with 75% or more reduction in the AK count in the Treatment Area as compared to baseline.
Time Frame: Baseline, Week 12
Measure: Number; unit: participants
Groups:
- Vehicle + BLUE Light Treatment: VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment at Visits 1 and 5. Subjects receiving VEH were considered a single treatment group.
  Vehicle PDT : Levulan Kerastick containing vehicle ingredients only.VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH were considered a single treatment group.
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants | 23 | 24 | 25 | 20 | 5

8. Secondary Outcome: Partial Clearance Rate
Description: proportion of subjects with 75% or more reduction in the AK count in the Treatment Area as compared to baseline.
Time Frame: Baseline Week 24
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants | 18 | 19 | 24 | 17 | 3

9. Secondary Outcome: AK Clearance Rate
Description: AK Clearance Rate (AKCR) for a subject is defined as:
  100% x [1 - (Number of AK lesions in the Treatment Area at follow-up visit/Number of AK lesions in the Treatment Area at Baseline)]
Time Frame: Baseline, Week 4
Measure: Median (Standard Deviation); unit: percent clearance
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
percent clearance | 40 (41.8) | 58.4 (34.8) | 54.5 (30.4) | 56.3 (54.3) | 0.0 (28.7)

10. Secondary Outcome: AK Clearance Rate
Description: as for outcome 9
Time Frame: Baseline, Week 8
Measure: Median (Standard Deviation); unit: percent clearance
Groups:
- Broad Area ALA 1-hour + BLUE Light Treatment: Broad Area ALA 1-hour incubation : 20% ALA, broad area, 1 hour incubation, prior to BLUE light treatment at Vist 1 and Visit 5
- Broad Area ALA 2-hour + BLUE Light Treatment: Broad Area ALA 2-hr incubation : 20% ALA broad area 2-hour incubation, prior to BLUE light treatment at Visit 1 and Visit 5
- Broad Area ALA 3-hour + BLUE Light Treatment: broad area ALA 3-hour incubation : 20% ALA broad area 3 hour incubation, prior to BLUE light treatment at Visit 1 and Visit 5
- Spot ALA 2-hour + BLUE Light Treatment: Spot application ALA 2 hour incubation : 20% ALA spot application 2 hour incubation, prior to BLUE light treatment at Visit 1 and Visit 5
- Vehicle + BLUE Light Treatment: VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment, at Visits 1 and 5. Subjects receiving VEH were considered a single treatment group.
  Vehicle PDT : Levulan Kerastick containing vehicle ingredients only.VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH were considered a single treatment group.
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
percent clearance | 35.7 (42.0) | 52.5 (37.2) | 57.1 (37.0) | 57.1 (43.8) | 5.7 (33.5)

11. Secondary Outcome: AK Clearance Rate
Description: as for outcome 9
Time Frame: Baseline, Week 12
Measure: Median (Standard Deviation); unit: percent clearance
Groups:
- Broad Area ALA 2-hour + BLUE Light Treatment: Broad Area ALA 2-hr incubation : 20% ALA broad area 2-hour incubation prior to BLUE light treatment at Vist 1 and Visit 5
- Broad Area ALA 3-hour + BLUE Light Treatment: broad area ALA 3-hour incubation : 20% ALA broad area 3 hour incubation, prior to BLUE light treatment at Vist 1 and Visit 5
- Spot ALA 2-hour + BLUE Light Treatment: Spot application ALA 2 hour incubation : 20% ALA spot application 2 hour incubation, prior to BLUE light treatment at Vist 1 and Visit 5
- Vehicle + BLUE Light Treatment: VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment at Vist 1 and Visit 5. Subjects receiving VEH were considered a single treatment group.
  Vehicle PDT : Levulan Kerastick containing vehicle ingredients only.VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH were considered a single treatment group.
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
percent clearance | 71.4 (34.8) | 73.6 (31.1) | 78.6 (30.5) | 68.3 (39.4) | 7.1 (44.3)

12. Secondary Outcome: AK Clearance Rate
Description: as for outcome 9
Time Frame: Baseline, Week 24
Measure: Median (Standard Deviation); unit: percent clearance
Groups:
- Broad Area ALA 2-hour + BLUE Light Treatment: Broad Area ALA 2-hr incubation : 20% ALA broad area 2-hour incubation, prior to BLUE light treatment at Vist 1 and Visit 5
- Vehicle + BLUE Light Treatment: VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment at Vist 1 and Visit 5 . Subjects receiving VEH were considered a single treatment group.
  Vehicle PDT : Levulan Kerastick containing vehicle ingredients only.VEH group was randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH were considered a single treatment group.
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
percent clearance | 66.7 (43.4) | 64.9 (36.3) | 75.0 (46.3) | 63.4 (44.3) | 14.3 (44.0)

13. Secondary Outcome: Subject Satisfaction Score
Description: 0 = no improvement or worsening (not satisfied at all)
  1. = slight improvement (slightly satisfied)
  2. = moderate improvement (moderately satisfied)
  3. = excellent improvement (very satisfied)
Time Frame: Week 24
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 46
participants
  3 = excellent improvement (very satisfied) | 20 | 21 | 20 | 20 | 7
  2 = moderate improvement (moderately satisfied) | 14 | 16 | 19 | 17 | 9
  1 = slight improvement (slightly satisfied) | 6 | 9 | 1 | 2 | 6
  0 = no improvement or worsening (not satisfied at | 7 | 2 | 4 | 7 | 24

14. Secondary Outcome: Hyperpigmentation at Baseline
Description: HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 12 | 8 | 17 | 14 | 11
  Grade 1 - Light | 23 | 24 | 23 | 21 | 27
  Grade 2 - Moderate/small | 12 | 14 | 6 | 9 | 7
  Grade 3 - Moderate/moderate | 0 | 2 | 1 | 2 | 1

15. Secondary Outcome: Hyperpigmentation at Visit 2
Description: as for outcome 14
Time Frame: 24-48 Hours after PDT #1
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 17 | 12 | 18 | 15 | 16
  Grade 1 - Light | 19 | 24 | 23 | 19 | 25
  Grade 2 - Moderate/small | 9 | 11 | 5 | 11 | 4
  Grade 3 - Moderate/moderate | 2 | 1 | 1 | 1 | 1

16. Secondary Outcome: Hyperpigmentation at Visit 3
Description: as for outcome 14
Time Frame: Week 2
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 16 | 10 | 20 | 16 | 15
  Grade 1 - Light | 18 | 27 | 21 | 23 | 24
  Grade 2 - Moderate/small | 12 | 10 | 5 | 7 | 4
  Grade 3 - Moderate/moderate | 1 | 1 | 1 | 0 | 2

17. Secondary Outcome: Hyperpigmentation at Visit 4
Description: as for outcome 14
Time Frame: Week 4
Population: Number of participants analyzed reflects ITT analysis of Tolerability Data, with no imputation techniques for missing data.
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 46 | 46 | 45
participants
  Grade 0 - None | 16 | 11 | 22 | 16 | 12
  Grade 1 - Light | 21 | 25 | 15 | 21 | 25
  Grade 2 - Moderate/small | 10 | 11 | 6 | 9 | 7
  Grade 3 - Moderate/moderate | 0 | 1 | 3 | 0 | 1

18. Secondary Outcome: Hyperpigmentation at Visit 5
Description: as for outcome 14
Time Frame: Week 8
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 45 | 46 | 44
participants
  Grade 0 - None | 16 | 11 | 17 | 14 | 11
  Grade 1 - Light | 19 | 26 | 20 | 23 | 25
  Grade 2 - Moderate/small | 12 | 10 | 7 | 8 | 6
  Grade 3 - Moderate/moderate | 0 | 1 | 1 | 1 | 2

19. Secondary Outcome: Hyperpigmentation at Visit 6
Description: as for outcome 14
Time Frame: Week 12
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 45 | 46 | 44
participants
  Grade 0 - None | 17 | 9 | 18 | 17 | 11
  Grade 1 - Light | 18 | 29 | 16 | 20 | 24
  Grade 2 - Moderate/small | 11 | 8 | 9 | 8 | 8
  Grade 3 - Moderate/moderate | 1 | 2 | 1 | 1 | 1

20. Secondary Outcome: Hyperpigmentation at Visit 7
Description: as for outcome 14
Time Frame: Week 24
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 46
participants
  Grade 0 - None | 16 | 9 | 20 | 18 | 13
  Grade 1 - Light | 23 | 27 | 19 | 21 | 25
  Grade 2 - Moderate/small | 7 | 10 | 4 | 6 | 7
  Grade 3 - Moderate/moderate | 0 | 2 | 1 | 1 | 1
  Grade 4 - Marked | 1 | 0 | 0 | 0 | 0

21. Secondary Outcome: Hypopigmentation at Baseline
Description: HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation Grade 4 = Marked hypopigmentation involving moderate or large sized areas
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 21 | 20 | 30 | 22 | 18
  Grade 1 - Light | 21 | 25 | 16 | 23 | 24
  Grade 2 - Moderate/small | 5 | 3 | 1 | 1 | 4

22. Secondary Outcome: Hypopigmentation at Visit 2
Description: as for outcome 21
Time Frame: 24-48 Hours after PDT #1
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 25 | 24 | 31 | 23 | 23
  Grade 1 - Light | 16 | 20 | 14 | 22 | 20
  Grade 2 - Moderate/small | 6 | 4 | 2 | 1 | 3

23. Secondary Outcome: Hypopigmentation at Visit 3
Description: as for outcome 21
Time Frame: Week 2
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 45
participants
  Grade 0 - None | 25 | 23 | 31 | 21 | 20
  Grade 1 - Light | 17 | 22 | 14 | 24 | 21
  Grade 2 - Moderate/small | 5 | 3 | 2 | 1 | 4

24. Secondary Outcome: Hypopigmentation at Visit 4
Description: as for outcome 21
Time Frame: Week 4
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 46 | 46 | 45
participants
  Grade - None | 25 | 20 | 29 | 19 | 19
  Grade 1 - Light | 17 | 21 | 16 | 26 | 22
  Grade 2 - Moderate/small | 5 | 1 | 0 | 1 | 4
  Grade 3 - Moderate/moderate | 0 | 0 | 1 | 0 | 0

25. Secondary Outcome: Hypopigmentation at Visit 5
Description: as for outcome 21
Time Frame: Week 8
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 45 | 46 | 44
participants
  Grade 0 - None | 23 | 19 | 28 | 17 | 18
  Grade 1 - Light | 21 | 26 | 17 | 25 | 23
  Grade 2 - Moderate/small | 3 | 3 | 0 | 4 | 3

26. Secondary Outcome: Hypopigmentation at Visit 6
Description: as for outcome 21
Time Frame: Week 12
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 44
participants
  Grade 0 - None | 23 | 20 | 26 | 19 | 15
  Grade 1 - Light | 21 | 26 | 18 | 20 | 26
  Grade 2 - Moderate/small | 3 | 2 | 0 | 6 | 3
  Grade 3 - Moderate/moderate | 0 | 0 | 0 | 1 | 0

27. Secondary Outcome: Hypopigmentation at Visit 7
Description: as for outcome 21
Time Frame: Week 24
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 46
participants
  Grade 0 - None | 22 | 18 | 28 | 20 | 17
  Grade 1 - Light | 22 | 27 | 15 | 24 | 25
  Grade 2 - Moderate/small | 3 | 3 | 1 | 2 | 4

28. Secondary Outcome: Erythema at Baseline
Description: Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 14 | 10 | 15 | 19 | 15
  Grade 1 - Minimal | 23 | 23 | 24 | 19 | 18
  Grade 2 Mild | 10 | 15 | 8 | 8 | 11
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 2

29. Secondary Outcome: Erythema Post-Light Treatment
Description: as for outcome 28
Time Frame: 5 minutes after PDT #1
Measure: Number; unit: participants
Groups:
- Broad Area ALA 1-hour + BLUE Light Treatment: Broad Area ALA 1-hour incubation : 20% ALA, broad area, 1 hour incubation, prior to BLUE light treatment at Visit 1 and Visit 5
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 2 | 0 | 0 | 0 | 4
  Grade 1 - Minimal | 8 | 4 | 5 | 9 | 25
  Grade 2 Mild | 19 | 16 | 13 | 18 | 14
  Grade 3 - Moderate | 16 | 26 | 22 | 18 | 3
  Grade 4 - Severe | 2 | 2 | 7 | 1 | 0

30. Secondary Outcome: Erythema at Visit 2
Description: as for outcome 28
Time Frame: 24-48 hours after PDT #1
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 2 | 0 | 1 | 0 | 13
  Grade 1 - Minimal | 8 | 3 | 4 | 11 | 17
  Grade 2 Mild | 10 | 14 | 12 | 9 | 14
  Grade 3 - Moderate | 25 | 23 | 18 | 24 | 2
  Grade 4 - Severe | 2 | 8 | 12 | 2 | 0

31. Secondary Outcome: Erythema at Visit 3
Description: as for outcome 28
Time Frame: Week 2
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 45
participants
  Grade 0 - None | 11 | 5 | 11 | 14 | 15
  Grade 1 - Minimal | 22 | 23 | 19 | 26 | 21
  Grade 2 Mild | 13 | 18 | 14 | 6 | 8
  Grade 3 - Moderate | 1 | 2 | 3 | 0 | 1
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Erythema at Visit 4
Description: as for outcome 28
Time Frame: Week 4
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 46 | 46 | 45
participants
  Grade 0 - None | 12 | 13 | 16 | 12 | 14
  Grade 1 - Minimal | 27 | 22 | 20 | 26 | 18
  Grade 2 Mild | 8 | 13 | 9 | 7 | 12
  Grade 3 - Moderate | 0 | 0 | 1 | 1 | 1
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

33. Secondary Outcome: Erythema at Visit 5 (Pre-drug)
Description: as for outcome 28
Time Frame: Week 8 pre-drug
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 45 | 46 | 44
participants
  Grade 0 - None | 13 | 15 | 17 | 21 | 12
  Grade 1 - Minimal | 25 | 17 | 22 | 19 | 20
  Grade 2 Mild | 9 | 16 | 5 | 6 | 10
  Grade 3 - Moderate | 0 | 0 | 1 | 0 | 2
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

34. Secondary Outcome: Erythema at Visit 5 (Post-light)
Description: as for outcome 28
Time Frame: Week 8 5 minutes post light treatment
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 41 | 37 | 31 | 41 | 44
participants
  Grade 0 - None | 1 | 0 | 1 | 0 | 4
  Grade 1 - Minimal | 8 | 5 | 7 | 9 | 28
  Grade 2 Mild | 19 | 10 | 7 | 19 | 7
  Grade 3 - Moderate | 12 | 19 | 16 | 13 | 5
  Grade 4 - Severe | 1 | 3 | 0 | 0 | 0

35. Secondary Outcome: Erythema at Visit 6
Description: as for outcome 28
Time Frame: Week 12
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 44
participants
  Grade 0 - None | 16 | 15 | 18 | 22 | 17
  Grade 1 - Minimal | 24 | 23 | 19 | 19 | 18
  Grade 2 Mild | 7 | 10 | 7 | 4 | 8
  Grade 3 - Moderate | 0 | 0 | 0 | 1 | 1
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: Erythema at Visit 7
Description: as for outcome 28
Time Frame: Week 24
Population: as for outcome 17
Measure: Number; unit: participants
Groups:
- Broad Area ALA 2-hour + BLUE Light Treatment at Visit 1 and Vi: Broad Area ALA 2-hr incubation : 20% ALA broad area 2-hour incubation, prior to BLUE light treatment at Visit 1 and Visit 5
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment at Visit 1 and Vi | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 46
participants
  Grade 0 - None | 20 | 16 | 19 | 27 | 21
  Grade 1 - Minimal | 19 | 20 | 20 | 15 | 16
  Grade 2 Mild | 7 | 12 | 5 | 4 | 7
  Grade 3 - Moderate | 1 | 0 | 0 | 0 | 2
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

37. Secondary Outcome: Edema at Baseline
Description: EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 0 | 0 | 1 | 0 | 0
  Grade 1 - Minimal | 0 | 0 | 0 | 0 | 0
  Grade 2 - Mild | 0 | 0 | 0 | 0 | 0
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

38. Secondary Outcome: Edema Post-Light Treatment
Description: as for outcome 37
Time Frame: 5 minutes after PDT #1
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 37 | 28 | 27 | 33 | 44
  Grade 1 - Minimal | 8 | 12 | 11 | 10 | 2
  Grade 2 - Mild | 2 | 7 | 3 | 3 | 0
  Grade 3 - Moderate | 0 | 1 | 6 | 0 | 0
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

39. Secondary Outcome: Edema at Visit 2
Description: as for outcome 37
Time Frame: 24-48 hours post PDT#1
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 32 | 31 | 26 | 27 | 44
  Grade 1 - Minimal | 8 | 10 | 10 | 13 | 2
  Grade 2 - Mild | 5 | 3 | 6 | 4 | 0
  Grade 3 - Moderate | 2 | 3 | 4 | 2 | 0
  Grade 4 - Severe | 0 | 1 | 1 | 0 | 0

40. Secondary Outcome: Edema at Visit 3
Description: as for outcome 37
Time Frame: Week 2
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 45
participants
  Grade 0 - None | 46 | 44 | 42 | 44 | 44
  Grade 1 - Minimal | 1 | 2 | 1 | 2 | 1
  Grade 2 - Mild | 0 | 2 | 4 | 0 | 0
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Edema at Visit 4
Description: as for outcome 37
Time Frame: Week 4
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 46 | 46 | 45
participants
  Grade 0 - None | 46 | 47 | 46 | 46 | 45
  Grade 1 - Minimal | 1 | 1 | 0 | 0 | 0
  Grade 2 - Mild | 0 | 0 | 0 | 0 | 0
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

42. Secondary Outcome: Edema at Visit 5 (Pre-drug)
Description: as for outcome 37
Time Frame: Week 8 pre-drug
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 45 | 46 | 44
participants
  Grade 0 - None | 47 | 48 | 45 | 46 | 44
  Grade 1 - Minimal | 0 | 0 | 0 | 0 | 0
  Grade 2 - Mild | 0 | 0 | 0 | 0 | 0
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

43. Secondary Outcome: Edema Post PDT #2
Description: as for outcome 37
Time Frame: 5 minutes post PDT #2
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 41 | 37 | 31 | 41 | 44
participants
  Grade 0 - None | 32 | 20 | 18 | 26 | 43
  Grade 1 - Minimal | 6 | 12 | 7 | 11 | 1
  Grade 2 - Mild | 2 | 4 | 3 | 4 | 0
  Grade 3 - Moderate | 1 | 1 | 3 | 0 | 0
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Edema at Week 12
Description: as for outcome 37
Time Frame: Week 12
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 44
participants
  Grade 0 - None | 47 | 48 | 43 | 46 | 44
  Grade 1 - Minimal | 0 | 0 | 1 | 0 | 0
  Grade 2 - Mild | 0 | 0 | 0 | 0 | 0
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

45. Secondary Outcome: Edema at Week 24
Description: as for outcome 37
Time Frame: Week 24
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 46
participants
  Grade 0 - None | 47 | 48 | 43 | 45 | 45
  Grade 1 - Minimal | 0 | 0 | 1 | 1 | 1
  Grade 2 - Mild | 0 | 0 | 0 | 0 | 0
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

46. Secondary Outcome: Stinging/Burning at Baseline
Description: STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable The most intense stinging/burning sensation during the 16 minute 40 second light treatment will be recorded.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 47 | 48 | 47 | 46 | 44
  Grade 1 - MInimal | 0 | 0 | 0 | 0 | 2
  Grade 2 - Moderate | 0 | 0 | 0 | 0 | 0
  Grade 3 - Severe | 0 | 0 | 0 | 0 | 0

47. Secondary Outcome: Stinging/Burning During Light Treatment
Description: as for outcome 46
Time Frame: During PDT #1 (most intense sensation)
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 2 | 1 | 0 | 3 | 35
  Grade 1 - MInimal | 15 | 9 | 10 | 16 | 11
  Grade 2 - Moderate | 23 | 29 | 22 | 19 | 6
  Grade 3 - Severe | 7 | 9 | 15 | 8 | 0

48. Secondary Outcome: Stinging/Burning Post Light-Treatment
Description: as for outcome 46
Time Frame: 5 minutes post PDT #1
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 8 | 5 | 1 | 8 | 40
  Grade 1 - MInimal | 29 | 17 | 19 | 25 | 6
  Grade 2 - Moderate | 8 | 25 | 19 | 13 | 0
  Grade 3 - Severe | 2 | 1 | 8 | 0 | 0

49. Secondary Outcome: Stinging/Burning at Visit 2
Description: as for outcome 46
Time Frame: 24-48 hours post PDT #1
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 25 | 23 | 20 | 35 | 41
  Grade 1 - MInimal | 18 | 20 | 17 | 10 | 4
  Grade 2 - Moderate | 4 | 4 | 7 | 1 | 1
  Grade 3 - Severe | 0 | 1 | 3 | 0 | 0

50. Secondary Outcome: Stinging/Burning at Visit 3
Description: as for outcome 46
Time Frame: Week 2
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 45
participants
  Grade 0 - None | 46 | 45 | 44 | 46 | 45
  Grade 1 - MInimal | 1 | 3 | 2 | 0 | 0
  Grade 2 - Moderate | 0 | 0 | 1 | 0 | 0
  Grade 3 - Severe | 0 | 0 | 0 | 0 | 0

51. Secondary Outcome: Stinging/Burning at Visit 4
Description: as for outcome 46
Time Frame: Week 4
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 46 | 46 | 44
participants
  Grade 0 - None | 45 | 47 | 46 | 46 | 44
  Grade 1 - MInimal | 2 | 1 | 0 | 0 | 0
  Grade 2 - Moderate | 0 | 0 | 0 | 0 | 1
  Grade 3 - Severe | 0 | 0 | 0 | 0 | 0

52. Secondary Outcome: Stinging/Burning at Visit 5 (Pre-drug)
Description: as for outcome 46
Time Frame: Week 8 prior to drug
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 45 | 46 | 44
participants
  Grade 0 - None | 47 | 48 | 45 | 45 | 42
  Grade 1 - MInimal | 0 | 0 | 0 | 1 | 2
  Grade 2 - Moderate | 0 | 0 | 0 | 0 | 0
  Grade 3 - Severe | 0 | 0 | 0 | 0 | 0

53. Secondary Outcome: Stinging/Burning at Visit 5 During PDT#2
Description: as for outcome 46
Time Frame: during PDT #2
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 41 | 37 | 31 | 41 | 44
participants
  Grade 0 - None | 4 | 1 | 0 | 4 | 28
  Grade 1 - MInimal | 20 | 11 | 7 | 23 | 16
  Grade 2 - Moderate | 15 | 20 | 16 | 13 | 0
  Grade 3 - Severe | 2 | 5 | 8 | 1 | 0

54. Secondary Outcome: Stinging/Burning at Visit 5 Post PDT#2
Description: as for outcome 46
Time Frame: 5 minutes post PDT #2
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 31 | 37 | 31 | 41 | 44
participants
  Grade 0 - None | 7 | 2 | 2 | 10 | 35
  Grade 1 - MInimal | 26 | 18 | 14 | 22 | 9
  Grade 2 - Moderate | 8 | 15 | 11 | 9 | 0
  Grade 3 - Severe | 0 | 2 | 4 | 0 | 0

55. Secondary Outcome: Stinging/Burning at Visit 6
Description: as for outcome 46
Time Frame: Week 12
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 44
participants
  Grade 0 - None | 47 | 48 | 44 | 44 | 43
  Grade 1 - MInimal | 0 | 0 | 0 | 2 | 1
  Grade 2 - Moderate | 0 | 0 | 0 | 0 | 0
  Grade 3 - Severe | 0 | 0 | 0 | 0 | 0

56. Secondary Outcome: Stinging/Burning at Visit 7
Description: as for outcome 46
Time Frame: Week 24
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 46
participants
  Grade 0 - None | 47 | 48 | 44 | 45 | 46
  Grade 1 - MInimal | 0 | 0 | 0 | 1 | 0
  Grade 2 - Moderate | 0 | 0 | 0 | 0 | 0
  Grade 3 - Severe | 0 | 0 | 0 | 0 | 0

57. Secondary Outcome: Scaling and Dryness at Baseline
Description: SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 25 | 24 | 26 | 29 | 16
  Grade 1 - Minimal | 16 | 19 | 17 | 15 | 21
  Grade 2 - Mild | 6 | 5 | 4 | 2 | 6
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 3
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

58. Secondary Outcome: Scaling and Dryness at Visit 2
Description: as for outcome 57
Time Frame: 24-48 hours after PDT #1
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 19 | 20 | 22 | 17 | 18
  Grade 1 - Minimal | 13 | 16 | 15 | 23 | 22
  Grade 2 - Mild | 10 | 8 | 4 | 6 | 6
  Grade 3 - Moderate | 5 | 4 | 5 | 0 | 0
  Grade 4 - Severe | 0 | 0 | 1 | 0 | 0

59. Secondary Outcome: Scaling and Dryness at Visit 3
Description: as for outcome 57
Time Frame: Week 2
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 22 | 21 | 20 | 27 | 19
  Grade 1 - Minimal | 17 | 15 | 16 | 16 | 20
  Grade 2 - Mild | 7 | 8 | 8 | 3 | 6
  Grade 3 - Moderate | 1 | 3 | 3 | 0 | 0
  Grade 4 - Severe | 0 | 1 | 0 | 0 | 0

60. Secondary Outcome: Scaling and Dryness at Visit 4
Description: as for outcome 57
Time Frame: Week 4
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 46 | 46 | 45
participants
  Grade 0 - None | 24 | 24 | 27 | 28 | 18
  Grade 1 - Minimal | 19 | 18 | 17 | 14 | 22
  Grade 2 - Mild | 3 | 6 | 1 | 4 | 4
  Grade 3 - Moderate | 1 | 0 | 1 | 0 | 1
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

61. Secondary Outcome: Scaling and Dryness at Visit 5
Description: as for outcome 57
Time Frame: Week 8
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 45 | 46 | 44
participants
  Grade 0 - None | 23 | 30 | 31 | 31 | 17
  Grade 1 - Minimal | 21 | 16 | 11 | 13 | 18
  Grade 2 - Mild | 3 | 2 | 3 | 2 | 9
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

62. Secondary Outcome: Scaling and Dryness at Visit 6
Description: as for outcome 57
Time Frame: Week 12
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 44
participants
  Grade 0 - None | 32 | 34 | 30 | 33 | 23
  Grade 1 - Minimal | 13 | 12 | 13 | 11 | 17
  Grade 2 - Mild | 2 | 2 | 0 | 2 | 4
  Grade 3 - Moderate | 0 | 0 | 1 | 0 | 0
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

63. Secondary Outcome: Scaling and Dryness at Visit 7
Description: as for outcome 57
Time Frame: Week 24
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 46
participants
  Grade 0 - None | 31 | 26 | 32 | 37 | 28
  Grade 1 - Minimal | 13 | 22 | 11 | 8 | 12
  Grade 2 - Mild | 3 | 0 | 1 | 1 | 5
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 1
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

64. Secondary Outcome: Oozing/Vesiculation/Crusting at Baseline
Description: OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 45 | 47 | 46 | 43 | 44
  Grade 1 - Minimal | 1 | 0 | 1 | 3 | 1
  Grade 2 - Mild | 1 | 1 | 0 | 0 | 1
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0

65. Secondary Outcome: Oozing/Vesiculation/Crusting at Visit 2
Description: as for outcome 64
Time Frame: 24-48 hours after PDT #1
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 46
participants
  Grade 0 - None | 43 | 39 | 34 | 34 | 43
  Grade 1 - Minimal | 2 | 4 | 5 | 9 | 2
  Grade 2 - Mild | 2 | 4 | 4 | 2 | 1
  Grade 3 - Moderate | 0 | 1 | 4 | 1 | 0
  Grade 4 - Severe | 0 | 0 | 0 | 0 | 0

66. Secondary Outcome: Oozing/Vesiculation/Crusting at Visit 3
Description: as for outcome 64
Time Frame: Week 2
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 45
participants
  Grade 0 - None | 45 | 42 | 45 | 45 | 45
  Grade 1 - Minimal | 1 | 5 | 1 | 0 | 0
  Grade 2 - Mild | 1 | 1 | 1 | 1 | 0
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0

67. Secondary Outcome: Oozing/Vesiculation/Crusting at Visit 4
Description: as for outcome 64
Time Frame: Week 4
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 46 | 46 | 45
participants
  Grade 0 - None | 46 | 45 | 46 | 46 | 45
  Grade 1 - Minimal | 1 | 3 | 0 | 0 | 0
  Grade 2 - Mild | 0 | 0 | 0 | 0 | 0
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0

68. Secondary Outcome: Oozing/Vesiculation/Crusting at Visit 5
Description: as for outcome 64
Time Frame: Week 8
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 45 | 46 | 44
participants
  Grade 0 - None | 47 | 47 | 45 | 44 | 42
  Grade 1 - Minimal | 0 | 1 | 0 | 2 | 1
  Grade 2 - Mild | 0 | 0 | 0 | 0 | 0
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 1

69. Secondary Outcome: Oozing/Vesiculation/Crusting at Visit 6
Description: as for outcome 64
Time Frame: Week 12
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 44
participants
  Grade 0 - None | 46 | 48 | 44 | 46 | 44
  Grade 1 - Minimal | 1 | 0 | 0 | 0 | 0
  Grade 2 - Mild | 0 | 0 | 0 | 0 | 0
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0

70. Secondary Outcome: Oozing/Vesiculation/Crusting at Visit 7
Description: as for outcome 64
Time Frame: Week 24
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Broad Area ALA 1-hour + BLUE Light Treatment | Broad Area ALA 2-hour + BLUE Light Treatment | Broad Area ALA 3-hour + BLUE Light Treatment | Spot ALA 2-hour + BLUE Light Treatment | Vehicle + BLUE Light Treatment
Number analyzed (Participants) | 47 | 48 | 44 | 46 | 46
participants
  Grade 0 - None | 47 | 48 | 44 | 45 | 46
  Grade 1 - Minimal | 0 | 0 | 0 | 1 | 0
  Grade 2 - Mild | 0 | 0 | 0 | 0 | 0
  Grade 3 - Moderate | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Broad Area ALA 1-hour: Broad Area ALA 1-hour incubation : 20% ALA, broad area, 1 hour incubation
- Broad Area ALA 2-hour: Broad Area ALA 2-hr incubation : 20% ALA broad area 2-hour incubation
- Broad Area ALA 3-hour: broad area ALA 3-hour incubation : 20% ALA broad area 3 hour incubation
- Spot ALA 2-hour: Spot application ALA 2 hour incubation : 20% ALA spot application 2 hour incubation
- Vehicle PDT: VEH group will be randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH will be considered a single treatment group.
  Vehicle PDT : Levulan Kerastick containing vehicle ingredients only.VEH group will be randomized (1:1:1:1) to be balanced for the four active groups; broad area application for 1, 2 or 3 hours or spot application for 2 hours prior to BLUE light treatment. Subjects receiving VEH will be considered a single treatment group.
Arm/Group | Broad Area ALA 1-hour | Broad Area ALA 2-hour | Broad Area ALA 3-hour | Spot ALA 2-hour | Vehicle PDT
Serious Adverse Events (participants affected / at risk) | 5/48 | 1/48 | 3/47 | 2/46 | 2/46
Other Adverse Events (participants affected / at risk) | 0/48 | 1/48 | 1/47 | 4/46 | 4/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Broad Area ALA 1-hour (N=48) | Broad Area ALA 2-hour (N=48) | Broad Area ALA 3-hour (N=47) | Spot ALA 2-hour (N=46) | Vehicle PDT (N=46)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
community-acquired pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
exacerbation of atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
splenectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Broad Area ALA 1-hour (N=48) | Broad Area ALA 2-hour (N=48) | Broad Area ALA 3-hour (N=47) | Spot ALA 2-hour (N=46) | Vehicle PDT (N=46)
squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of results from multi-center trial will be made by the Sponsor. If publication is not submitted within 12 months after conclusion of the study, the PI may publish the results from the site individually, subject to compliance with the other terms of the clinical trial agreement, including a requirement that the PI provide a draft of the publication for the sponsor's review 60 days before publication so that sponsor can review the publication for confidential information.